CLINICAL TRIAL: NCT06001125
Title: A Study to Evaluate the Efficacy and Safety of Methotrexate in Immune Related Arthritis or Arthralgias
Brief Title: Methotrexate for Immune Related Arthritis or Arthralgias (IMPACT 2.1)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Challenges in meeting the enrollment target
Sponsor: AHS Cancer Control Alberta (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IIT-0029
Record Dates: First submitted 2023-08-04; First posted 2023-08-21 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2026-01

CONDITIONS: Arthritis; Arthralgia
MeSH Terms: conditions — Arthritis; Arthralgia | interventions — Methotrexate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single Arm (Experimental): Methotrexate 20 mg PO weekly for 12 weeks.
  Folic acid 1mg PO daily for as long as Methotrexate is given.
  Prednisone starting at 20 mg PO daily for 8 weeks tapering dose.
  Interventions: Drug: Methotrexate

INTERVENTIONS:
Drug: Methotrexate — Methotrexate 20 mg PO weekly

SUMMARY:
Many people develop joint pain, stiffness and swelling due to their cancer treatment that targets the immune system.

The severity of symptoms ranges from mild to debilitating and sometimes requires delaying or stopping cancer treatment.

The usual plan is to discontinue cancer treatment and give relatively high doses of a medication called prednisone (a steroid, which is an anti-inflammatory medication which may suppress the immune system), with a gradual lowering of the dose over several weeks.

While this can be effective, prednisone can cause several side effects, and it is not known if this is the best or safest treatment.

Hydroxychloroquine is a medication being studied on IMPACT 2.0 on participants who develop inflammatory joint pain while taking cancer treatments that affect their immune system. It is possible that the hydroxychloroquine treatment may not work well on some participants on IMPACT 2.0. Hydroxychloroquine is also given as standard of care to participants with this type of inflammatory joint pain.

The goal of this study is to learn how well methotrexate is at treating inflammatory joint pain in participants from IMPACT 2.0 that don't do well on treatment with hydroxychloroquine and in patients given hydroxychloroquine as standard of care to treat this type of inflammatory joint pain caused by taking cancer treatments which target their immune system.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who were previously on hydroxychloroquine treatment as standard of care therapy or enrolled in IMPACT 2.0 who develop recurrent grade ≥ 2 irAA, or who remain on glucocorticoids for irAA at 3 months will be eligible for this trial.
2. Patients must be 18 years of age, or older.
3. Patients must be capable of providing consent to enrolment and treatment.
4. Patients with a performance status of ECOG 0-2 will be eligible for enrolment.
5. Patients with histologically confirmed cancer receiving anti-PD1 or anti-PDL1 monoclonal antibody ICI therapy, either alone or in combination with anti-CTLA4 monoclonal antibody ICI therapy who develop CTCAEv5.0 grade ≥2 arthritis or arthralgia that has developed on, or after, ICI therapy and is felt to be treatment related (irAA).
6. Adequate hematologic parameters defined by the following laboratory parameters:

   * Hgb >100 g/L
   * Platelets>150 x 109/L
   * WBC>Lower limit of normal
7. Adequate hepatic and renal function defined by the following laboratory parameters:

   * AST, ALT, bilirubin and alkaline phosphatase within normal range,
   * Serum creatinine ≤ upper limit of institutional normal OR calculated creatinine clearance of ≥ 60 mL/min using the Cockcroft-Gault formula.
   * Patients with an elevated bilirubin, but confirmed to have Gilbert's disease will be eligible
8. Women of childbearing potential (WOCBP) must have a negative serum (or urine) pregnancy test at the time of screening. WOCBP is defined as any female who has experienced menarche and who has not undergone surgical sterilization (hysterectomy or bilateral oophorectomy or bilateral salpingectomy) and is not postmenopausal. Menopause is defined as 12 months of amenorrhea in a woman over age 45 years in the absence of other biological or physiological causes. In addition, females under the age of 55 years must have a serum follicle stimulating hormone, (FSH) level > 40 mIU/mL to confirm menopause.
9. Patients of childbearing/reproductive potential should use highly effective birth control methods, during the study treatment period and for a period of 6 months after the last dose of study drug. A highly effective method of birth control is defined as those that result in low failure rate (i.e., less than 1% per year) when used consistently and correctly. These may include hormonal contraceptives (e.g., combined oral contraceptives, patch, vaginal ring, injectables, and implants); intrauterine device (IUD) or intrauterine system (IUS); vasectomy and tubal ligation. Double-barrier methods may be acceptable in circumstances when highly effective methods cannot be implemented (e.g., male condom with diaphragm, male condom with cervical cap). Note: Contraceptive requirements for the oncology regiments will apply, if they are more stringent than those for this trial. Abstinence is acceptable if this is established and preferred contraception for the patient.
10. Female patients who are breast-feeding should discontinue nursing prior to the first dose of study treatment and until 6 months after the last dose of study drug.
11. Male patients should agree to not donate sperm during the study and for a period of at least 6 months after last dose of study drug.
12. Absence of any condition hampering compliance with the study protocol and follow- up schedule; those conditions should be discussed with the patient before registration in the trial.

Exclusion Criteria:

1. History of inflammatory arthritis, including, but not limited to: Rheumatoid arthritis, systemic lupus erythematosus, Sjogren's syndrome, Ankylosing spondylitis or other chronic inflammatory arthritis. Note: Patients with a known history of stable osteoarthritis will not be excluded.
2. Patients with an indication for systemic immunosuppressive medications or corticosteroids. Patients with CTCAEv5.0 grade ≥2 irAE's other than irAA (ie. colitis, pneumonitis, rash, etc) are not eligible for trial, with the exception of endocrinopathies that are being treated with hormone replacement alone and not systemic immunosuppressive medications or corticosteroids.
3. Patients with G6PD deficiency, porphyria or psoriasis.
4. Clinically significant (i.e., active) cardiovascular disease: cerebral vascular accident/stroke (< 6 months prior to enrollment), myocardial infarction (< 6 months prior to enrollment), unstable angina, congestive heart failure (≥ New York Heart Association Classification Class II), or serious cardiac arrhythmia requiring medication.
5. Diagnosis of immunodeficiency.
6. Diagnosis of untreated hepatitis B and C.
7. Current use of immunosuppressive medication, EXCEPT for the following: prednisone and hydroxychloroquine per IMPACT 2.0 protocol or standard of care.
8. Known prior severe hypersensitivity to investigational product or any component in its formulations, including known severe hypersensitivity reactions to monoclonal antibodies (CTCAEv5.0 Grade ≥ 3).
9. Excessive alcohol intake defined as greater than 7 units per week.
10. Other severe acute or chronic medical conditions including inflammatory bowel disease, immune pneumonitis, pulmonary fibrosis or psychiatric conditions including recent (within the past year) or active suicidal ideation or behavior; or laboratory abnormalities (see parameters in inclusion criteria) that may increase the risk associated with study participation or study treatment administration or may interfere with the interpretation of study results and, in the judgment of the investigator, would make the patient inappropriate for entry into this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2024-08-12 (Actual); Primary Completion 2025-06-17 (Actual); Study Completion 2025-10-07 (Actual)

PRIMARY OUTCOMES:
Discontinuation of Prednisone | 12 weeks
  Proportion of patients who were able to discontinue prednisone by 12 weeks without recurrence of grade 2 or higher irAA.

SECONDARY OUTCOMES:
Total Steroid Usage | 12 weeks
  The total cumulative dose of prednisone measured in mg used by the participant. If corticosteroids other than prednisone are used, their equivalent dosage in mg of prednisone will be calculated and used for this analysis.
Development of Immune Related Adverse Events (irAEs) Other Than irAA | 12 weeks
  Defined as the emergence of adverse events that were not present at study baseline that are deemed by the investigator to be related to prior use of immune checkpoint inhibitors. Causality will be investigator assessed and graded according to CTCAEv5.0
Adverse Events | 12 weeks
  The emergence of new or worsening baseline symptoms, physical findings, or laboratory/imaging abnormalities. Causality to study treatment, immune checkpoint inhibitors, or underlying disease status will be investigator assessed and graded according to CTCAEv5.0.
Re-initiation of Immune Checkpoint Inhibitor Therapy | 12 weeks
  The proportion of participants in each study arm that are re-treated with an immune checkpoint inhibitor.
Progression Free Survival | Time Frame: Total study observation period (3 years)
  The time elapsed between recruitment and tumor progression (radiographically or clinically) or death from any cause.

OTHER OUTCOMES:
Musculoskeletal Ultrasound of Symptomatic Joints | Performed at baseline and Week 13 Day1 (to align with 12- month MSK Ultrasound of IMPACT 2.0). Analysis will be done to compare baseline to Wk13D1.
  Ultrasounds assessment of symptomatic joints identified through clinical examination, will be performed and severity of joint inflammation will be assessed.
RAPID 3 Questionnaire | Performed at screening, baseline, Week 3 Day 1, Week 5 Day 1, Week 7 Day 1, Week 9 Day 1, Week 11 Day 1, Week 13 Day 1, and at 6 and 12 month follow up.
  Patient reported outcomes (PROs) are an important and clinically relevant endpoint in clinical trials. The RAPID 3 Questionnaire is a brief, easy to complete questionnaire that provides an assessment of physical function, pain, and global health. It is a validated tool in rheumatoid arthritis. The investigators plan to monitor changes in RAPID 3 score over time.
Bone Turnover Markers | Collected at baseline, Week 13 Day 1
  Corticosteroids are known to promote loss of bone mineral density and predispose to osteoporosis.
T-cell phenotyping (peripheral blood monocytes) and T-cell Receptor Sequencing | Collected at baseline and at end of treatment (Week 13)
  T cell function is essential to the anti-cancer effect of ICI's. The investigators intend to collect PBMC's and perform T-cell phenotying and T-cell receptor sequencing and correlate this with irAE and cancer outcomes.
Immunophenotyping | Collected at baseline and at end of treatment (Week 13)
  Immunophenotyping of regulatory T cells, expression of co-inhibitory receptors and ligands on T and the expression of T cells activation markers and the frequency of CD71+ erythroid cells because Methotrexate can impact the erythropoiesis.
Cytokine Profile | Collected at baseline and at end of treatment (Week 13)
  The cytokine profiles of different types of inflammatory arthritis are distinct and may predict response to difference types of treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Kolinsky, Principal Investigator — AHS-CCI
Locations (1):
- Cross Cancer Institute, Edmonton, Canada